CLINICAL TRIAL: NCT06585735
Title: Impact of Proteolytic Enzyme Fortified Protein Supplement in Patients With Chronic Pancreatitis.
Brief Title: Proteolytic Enzyme Fortified Protein Supplement in Chronic Pancreatitis.
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Asian Institute of Gastroenterology, India (Other)
Responsible Party: Principal Investigator, Rupjyoti Talukdar, Rupjyoti Talukdar, Asian Institute of Gastroenterology, India
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PEFP2024
Record Dates: First submitted 2024-08-18; First posted 2024-09-05 (Actual); Last update posted 2024-09-05 (Actual); Status verified 2024-09

CONDITIONS: Chronic Pancreatitis; Malnutrition
Keywords: chronic pancreatitis; malnutrition; enzyme fortified protein supplementation; randomised controlled trial
MeSH Terms: conditions — Pancreatitis, Chronic; Malnutrition

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Experimental): Group I receive 15 gms of Protein supplements (proteolytic enzyme with 70000 Hb unit tyrosine [HUT] fortified with 15 gms of whey protein), given daily for 6 weeks.
  Interventions: Dietary Supplement: Proteolytic enzyme fortified protein supplement
- Group B (Active Comparator): Group II will receive equivalent dose of plain protein supplement without proteolytic enzyme, given daily for 6 weeks.
  Interventions: Dietary Supplement: Proteolytic enzyme fortified protein supplement

INTERVENTIONS:
Dietary Supplement: Proteolytic enzyme fortified protein supplement — Group I receive Enzotein 15 gms (proteolytic enzyme with 70000 Hb unit tyrosine (HUT) fortified with 15 gms of whey protein), given for 6 weeks. Enzotein will be provided by (Mylin Biotech India Ltd.)

SUMMARY:
A complex disease, Chronic Pancreatitis (CP) is caused by a wide range of factors, including smoking, alcoholism, autoimmune disorders, and obstruction of the major pancreatic duct. In patients who are genetically susceptible to the condition, these factors can result in damage to the acinar, ductal, and islet cells, as well as persistent inflammatory infiltration and fibrosis. Malnutrition is an ongoing concern for persons with CP, even though pain is the primary symptom in most cases. Complications that commonly arise during the disease's natural history include exocrine and endocrine pancreatic insufficiency and local changes (such as pseudocyst, biliary and duodenal blockage, splenic and portal vein thrombosis, and pancreatic cancer). Consequently, CP mortality is higher than that of the general population.

DETAILED DESCRIPTION:
Maldigestion due to pancreatic exocrine insufficiency (PEI) and food avoidance (because by pain) are two physical causes of malnutrition1. Delayed gastric emptying leads to nausea, vomiting, and poor oral intake due to duodenal stenosis or extrinsic compressions of the stomach or duodenum from pseudocysts1. Chronic pancreatitis can be difficult to manage nutritionally, but there are number of different approaches to help with a customized treatment plan for each patient. Patients require comprehensive nutrition care due to the possible combination of malnutrition and insufficient calorie intake. Estimated nutritional requirements are 1.2 to 1.5 g/kg protein and 25 to 35 kcal/kg energy12-14. The use of estimated weight-based nutritional requirements raises concerns because it does not account for malabsorption. It is unclear from the scant studies in this area whether the nutritional deficiency results from higher energy expenditure, impaired nutrient absorption, or a combination of the two15.

According to international guidelines, all patients should have a screening for malnutrition within 24 hours of being admitted to the hospital, and those who are at risk ought to receive appropriate nutritional therapies16,17. The ongoing disease process in CP increases the requirement for nutrition. Most CP patients can be treated with regular diet combined with exogenous pancreatic enzyme supplements. 10% to 15% of patients usually need oral nutrition supplements (this can be higher in clinical practice), and 5% of patients need tube feeding.

Oral dietary supplements are widely accessible and are chosen based on the specific requirements of each patient. It has been proposed that people with chronic pancreatitis benefit from the use of oral elemental supplements. Oral elemental supplements have been linked to improvements in nutrition indices and a significant decrease in pain levels18,19. Ito et al. showed that two patients with calcified chronic pancreatitis experienced significant pain reduction when they consumed an elemental diet orally without the need for tube feeding20. In addition, Shea et al. examined the benefits of an oral peptide-based diet containing medium-chain triglycerides (MCT) on eight individuals with chronic pancreatitis, demonstrating improvements in pain management21.

The current investigator initiated study, we hypothesize that pre-digested proteins could improve the intestinal absorption. With this premise, we aim to investigate the role of proteolytic enzyme fortified protein supplementation on the nutritional status of patients with chronic pancreatitis.

ELIGIBILITY:
Inclusion Criteria:

1. Patients diagnosed with Chronic pancreatitis and on PERT.
2. Patient who has given consent for the study.
3. Participants who are greater 18yrs of age
4. Patients on oral diet
5. BMI less than ≤ 20kgs/m2

Exclusion Criteria:

1. Patients with hemodynamic instability.
2. Patients with history of GI surgeries.
3. Patients on immunosuppressants
4. Patients having other malignancies.
5. Participants who are allergic/ intolerance to any of the ingredients in the supplement
6. Patients on enteral feeding or in combination with parenteral nutrition

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-09-01 (Estimated); Primary Completion 2025-03-31 (Estimated); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
Weight gain | 6 weeks
  Improvement in body weight at least by 10% of the original weight.

SECONDARY OUTCOMES:
Improvement in body composition | 6 weeks
  Change in composition in medical body composition analyser (mBCA) test
Improvement in body function 1 | 6 weeks
  Muscle strength will be assessed by Jamar Hand grip Dynamometer at baseline and at the end of 6 weeks.
Improvement in body function 2 | 6 weeks
  Muscle function will be assessed by SARC-F questionnaire at baseline and at the end of the 6 weeks
Improvement in body function 3 | 6 weeks
  Muscle performance will be assessed using a 6-minute walk test at baseline and at the end of the 6 weeks
Improvement in pain | 6 weeks
  Improvement in pain (VAS 0-10)

CONTACTS AND LOCATIONS:
Overall Officials: Rupyoti Talukdar, MD, Principal Investigator — Director, Pancreatology
Locations (1):
- Asian Institute of Gastroenterology Hospitals, Hyderabad, Telangana, India

IPD SHARING:
Plan to Share IPD: Undecided